CLINICAL TRIAL: NCT03936530
Title: Infrapyloric (No.206) and Greater Curvature (No.204) Lymph Node Metastasis in Adenocarcinoma Located at Hepatic Flexure and Right Half of Transverse Colon
Brief Title: Infrapyloric and Greater Curvature Lymph Node Metastasis in Colon Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Shanghai Minimally Invasive Surgery Center (Other)
Responsible Party: Sponsor
Other Study IDs: MISC- Infrapyloric LNM
Record Dates: First submitted 2019-05-02; First posted 2019-05-03 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Colorectal Neoplasm
Keywords: colon adenocarcinoma; lymph node metastasis; right hemi-colectomy
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The infrapyloric (No.206) and greater curvature (No.204) lymph node metastasis in adenocarcinoma located at hepatic flexure and right half of transverse colon has not been well discribed and analysed. The aim of this study is to assess the rate of this lymph node metastasis and to reveal its prognostic value for colon cancer located at hepatic flexure and right half of transverse colon. Meanwhile, we can evaluate the safety and feasibility of this extented lymphadenectomy in right hemi-colectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* American Society of Anesthesiologists (ASA) score I to III
* A biopsy proven histological diagnosis of colorectal carcinoma
* tumor located at hepatic flexure and right half of transverse colon
* Undergoing right hemi-colectomy with extented lymphadenectomy of infrapyloric (No.206) and greater curvature (No.204) lymph node
* Preoperative staging cT2-4aN0M0 or cTanyN+M0
* Willing to participate and informed consent signed

Exclusion Criteria:

* Pregnant or lactating women
* Synchronous colorectal carcinoma
* History of colorectal cancer or other malignant tumors
* Clinical evidence of metastasis
* Preoperative staging cT1N0 or cT4bNany
* Emergency procedure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in Shanghai Minimally Invasive Surgery Center
Sampling Method: Non-Probability Sample
Enrollment: 432 (Actual)
Dates: Start 2019-10-20 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
metastasis rate | an average of 1 year
  metastasis rate of infrapyloric (No.206) and greater curvature (No.204) lymph node

SECONDARY OUTCOMES:
lymphadenectomy time | an average of 1 year
  time of lymphadenectomy of infrapyloric (No.206) and greater curvature (No.204) lymph node
intraoperative complication | an average of 1 year
  intraoperative complication
postoperative complication | an average of 1 year
  postoperative complication
3-year DFS | an average of 3 years
  3-year disease free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Yalikun A, Cai Z, Hong HJ, Dai K, Li S, Kwan W, Ma J, Feng B, Lu A, Zheng M, Zang L. Infrapyloric (No. 206) and greater curvature (No. 204) lymph node metastasis in adenocarcinoma located in the right half of the transverse colon (InCLART Study): protocol for a multicentre prospective observational study. BMJ Open. 2023 Feb 21;13(2):e066981. doi: 10.1136/bmjopen-2022-066981. PMID 36810166